CLINICAL TRIAL: NCT04667780
Title: Study to Investigate the Treatment Effect of Colchicine in Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ayub Teaching Hospital (Other)
Collaborators: Universidad de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATH/IRB/Colchicine/25.11.2020
Record Dates: First submitted 2020-12-11; First posted 2020-12-16 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Phase III, prospective, randomized, controlled, open-label and pragmatic trial, comparing the administration of Colchicine plus standard treatment vs. standard therapy, in hospitalized patients with COVID-19, within the first 48 hours, and no severity criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): This arm will receive Standard COVID-19 care + Colchicine
  The Colchicine treatment includes an initial dose of 1.5 mg (1 mg and 0.5 mg two hours after), followed by 0.5 mg every 12 hours during the next 7 days and 0.5 mg every 24 hours until the completion of 14 days of total treatment. In patients receiving ritonavir or lopinavir or with reduced renal clearance (<50 ml/min/1.37m2), weight <70 kg or age >75 years old, the dose will be adjusted to the half.
  Interventions: Drug: Colchicine; Drug: Standard COVID-19 care
- Control - Standard COVID-19 care (Other): This arm will receive standard COVID-19 care as per the hospital guidelines.
  Interventions: Drug: Standard COVID-19 care

INTERVENTIONS:
Drug: Colchicine — Colchicine tablet 0.5 mg
  Arms: Colchicine
Drug: Standard COVID-19 care — As per the hospital guidelines

SUMMARY:
COVID-19 is associated with a cytokine storm that leads to respiratory distress, multiorgan failure and elevated mortality. Oral Colchicine exhibits high anti-inflammatory capacity attributed to the inhibition of microtubules polymerization, inflammasome and production of IL-1β and IL-6, which could prevent the inflammatory storm in COVID-19 patients at risk. The investigators present a randomized, controlled, open-labeled, and pragmatic clinical trial to study the treatment effect of Colchicine in COVID-19 patients requiring hospitalization, but no intensive care yet. Colchicine will be started within the first 48 hours and continue for 14 days using a descending dose. The benefits will be studied in terms of clinical evolution (WHO 7-point scale) and IL-6 levels, as well as other clinical and biochemical secondary end-points. In the case of positive results, the clinical impact would be relevant given that this oral medication is affordable and widely accessible which would help to prevent the inflammatory complications associated with COVID-19.

DETAILED DESCRIPTION:
This is a Phase III, prospective, pragmatic, randomized, controlled and open-label trial, comparing standard of care vs. standard of care plus COLCHICINE for 14 days, in patients hospitalized due to COVID-19 and confirmed infection by SARS-CoV-2, within the first 48 hours after the hospital admission. Patients meeting severity criteria will be excluded, defined as established limitation of therapeutic effort or need for invasive mechanical ventilation at the time of inclusion. The Colchicine treatment includes an initial dose of 1.5 mg (1 mg and 0.5 mg two hours after), followed by 0.5 mg every 12 hours during the next 7 days and 0.5 mg every 24 hours until the completion of 14 days of total treatment. In patients receiving ritonavir or lopinavir or with reduced renal clearance (<50 ml/min/1.37m2), weight <70 kg or age >75 years old, the dose will be adjusted to the half.

Patients meeting all the inclusion criteria and none of the exclusion ones (see below), after signing the informed consent, will be centrally randomized to "Colchicine" or "Control" group. Patients in both groups will receive the standard therapy for COVID-19 as per the hospital protocols. Randomization will be controlled by: age, sex, time from initiation of symptoms, cardiovascular disease, the 7 point WHO and levels of C-reactive protein, ferritin, D-dimer, IL-6 and lymphocyte levels.

ELIGIBILITY:
Inclusion Criteria:

1. SARS-CoV-2 infection confirmed by PCR.
2. Admitted in the hospital in the previous 48 hours, with clinical status 3, 4 or 5 of WHO classification.
3. Age above 18 years old.
4. Informed written consent.

Exclusion Criteria:

1. Invasive mechanical ventilation needed.
2. Established limitation of the therapeutic effort
3. Inflammatory bowel disease (IBD: Chron Syndrome or Ulcerative colitis), chronic diarrhea or malabsorption.
4. Previous neuromuscular disease.
5. Other disease with an estimated vital prognosis under 1 year.
6. Severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2)
7. Medical records of cirrhosis, active chronic hepatitis or severe hepatic disease defined by GOT or GPT levels three times above the normal upper limit.
8. Patients with previous colchicine treatment for other diseases (mainly chronic prescriptions for familial Mediterranean fever or gout). Clearance period will not be required for patients treated with colchicine who stopped the treatment before the randomization.
9. Patients with history of allergic reaction or significant sensitivity to colchicine.
10. Treatment with immunosuppressive agents, corticoids or interleukine-1 antagonists for 6 months before inclusion.
11. Pregnant or breastfeeding female, confirmed by a positive result in the human chorionic gonadotropin (hCG) test.
12. Fertile woman, or post-menopausal during less than one year and non-surgically sterilized. Women of fertile age may be included if using at least one contraceptive method and preferably two complementary contraceptive methods.
13. Use of other investigational drugs in the moment of inclusion, or during 30 days previous to inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Changes in the patients' clinical status through the 7 points ordinal scale WHO R&D Blueprint expert group | up to 14 days
  Improvement in the clinical evolution of patients
Changes in IL-6 concentrations | up to 14 days
  Improvement in cytokine level

SECONDARY OUTCOMES:
Improvement in the clinical status | up to 14 days
  time needed to reduce at least 2 points in the 7-point Ordinal Scale for Clinical Improvement by WHO R&D Blueprint expert group (0-7)
Changes in the score for the Sequential Organ Failure Assessment (SOFA score) | up to 14 days
  Sequential Organ Failure Assessment (SOFA score) (0-14)
Changes in the punctuation in the National Early Warning Score | up to 14 days
  National Early Warning Score (NEWS scale)
Number of days with invasive mechanical ventilation | up to 14 days
Number of days with high flow oxygen therapy | up to 14 days
Changes in other inflammatory markers | up to 14 days
  C-reactive protein
Changes in severity markers | up to 14 days
  D-dimer
Changes in severity markers | up to 14 days
  Leukocytes
Changes in severity markers | up to 14 days
  Lymphocytes
Changes in severity markers | up to 14 days
  Platelets
Changes in severity markers | up to 14 days
  LDH
Changes in severity markers | up to 14 days
  Ferritin
Changes in myocardial damage | up to 14 days
  myocardial stress markers hsTnT
Changes in myocardial damage | up to 14 days
  myocardial stress markers NT-proBNP
Time until reaching a virus negative status | up to 14 days
  RT-PCR assay
Length of hospital stay | up to 14 days
  Length of hospital stay
Number of days in the intensive care unit. | up to 14 days
  Number of days in the intensive care unit.
Mortality | up to 14 days
  Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Ayub Teaching Hospital, Abbottabad, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deftereos SG, Giannopoulos G, Vrachatis DA, Siasos GD, Giotaki SG, Gargalianos P, Metallidis S, Sianos G, Baltagiannis S, Panagopoulos P, Dolianitis K, Randou E, Syrigos K, Kotanidou A, Koulouris NG, Milionis H, Sipsas N, Gogos C, Tsoukalas G, Olympios CD, Tsagalou E, Migdalis I, Gerakari S, Angelidis C, Alexopoulos D, Davlouros P, Hahalis G, Kanonidis I, Katritsis D, Kolettis T, Manolis AS, Michalis L, Naka KK, Pyrgakis VN, Toutouzas KP, Triposkiadis F, Tsioufis K, Vavouranakis E, Martinez-Dolz L, Reimers B, Stefanini GG, Cleman M, Goudevenos J, Tsiodras S, Tousoulis D, Iliodromitis E, Mehran R, Dangas G, Stefanadis C; GRECCO-19 investigators. Effect of Colchicine vs Standard Care on Cardiac and Inflammatory Biomarkers and Clinical Outcomes in Patients Hospitalized With Coronavirus Disease 2019: The GRECCO-19 Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e2013136. doi: 10.1001/jamanetworkopen.2020.13136. PMID 32579195
- [Background] Scarsi M, Piantoni S, Colombo E, Airo P, Richini D, Miclini M, Bertasi V, Bianchi M, Bottone D, Civelli P, Cotelli MS, Damiolini E, Galbassini G, Gatta D, Ghirardelli ML, Magri R, Malamani P, Mendeni M, Molinari S, Morotti A, Salada L, Turla M, Vender A, Tincani A, Brucato A, Franceschini F, Furloni R, Andreoli L. Association between treatment with colchicine and improved survival in a single-centre cohort of adult hospitalised patients with COVID-19 pneumonia and acute respiratory distress syndrome. Ann Rheum Dis. 2020 Oct;79(10):1286-1289. doi: 10.1136/annrheumdis-2020-217712. Epub 2020 Jul 30. PMID 32732245